CLINICAL TRIAL: NCT04638595
Title: Pediatric Normative Movement Analysis Data Collection
Status: Completed | Type: Observational
Sponsor: MultiCare Health System Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Normative Data Study
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normative: 50 neurotypical pediatric subjects
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — This project seeks to recruit 25 male and 25 female typically developing children between the ages of 3 and 18 years of age. Non-invasive measurements of movement patterns will be collected during common activities of daily living over a single data collection session.

SUMMARY:
The objective of this project is to collect baseline data from a normative population of children that gender and age matches the population of patients expected to be treated by Mary Bridge Children's Therapy Services and seen in the Research and Movement Laboratory. This project seeks to recruit 25 male and 25 female typically developing children between the ages of 3 and 18 years of age. Non-invasive measurements of movement patterns will be collected during common activities of daily living over a single data collection session.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3-18 years
* Ambulate independently and without the use of assistive devices
* Perform activities of daily living without physical assistance
* Tolerate adhesive markers placed on skin and clothing
* Willing and interested in participating

Exclusion Criteria:

* Neuromuscular disorders such as cerebral palsy, muscular dystrophy, myotonic dystrophy, spinal muscular atrophy, peripheral neuropathy, or other generalized muscle and/or nerve issues
* Evidence of developmental delays, muscle weakness, decreased muscle tone, joint stiffness, muscle or bone deformity
* Currently using or has a history of using assistive technology devices, bracing/orthoses, manual or powered mobility equipment
* Was born pre-term
* Currently or has a history of taking medication or pharmaceutical treatment related to musculoskeletal side-effects/scenario/diagnosis

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A group of 50 neurotypical pediatric subjects will be recruited for this data collection. Children will be assigned to 1 of 5 age groupings (3-5, 6-8, 9-11, 12-14, 15-18), with an equal amount of male/female in each.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Create normative baseline data for typically developing children | 1 year
  Establishing a baseline of pediatric biomechanics is an important step in performing the best possible analyses for our patients. Normative data provides that baseline, and provides the data to explore links within the dense, interconnected behavior of human motion.

CONTACTS AND LOCATIONS:
Locations (1):
- Mary Bridge Children's Therapy Unit, Puyallup, Washington, United States

IPD SHARING:
Plan to Share IPD: No